CLINICAL TRIAL: NCT02143323
Title: A Clinical Study to Evaluate the Effect of Glutathion S-transferase Polymorphism on Pharmacokinetics/Pharmacodynamics After Multiple Administration of Amoxicillin/Clavulanate and Explore Biomarkers for Drug-induced Liver Injury (DILI)
Brief Title: A Clinical Study to Explore Biomarkers for Drug-induced Liver Injury (DILI)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, In-Jin Jang, MD, PhD, Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DILI_Healthy
Record Dates: First submitted 2014-01-18; First posted 2014-05-21 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
Keywords: GST, DILI, biomarker
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury | interventions — Amoxicillin-Potassium Clavulanate Combination; BID protein, human; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Glutathione S-Transferase Theta1(GSTT1)/Mu1(GSTM1) wild/wild (Active Comparator): Augmentin tablet
  Interventions: Drug: Augmentin tablet
- GSTT1/GSTM1 wild/null type (Active Comparator): Augmentin tablet
  Interventions: Drug: Augmentin tablet
- GSTT1/GSTM1 null/wild type (Active Comparator): Augmentin tablet
  Interventions: Drug: Augmentin tablet
- GSTT1/GSTM1 null/null type (Active Comparator): Augmentin tablet
  Interventions: Drug: Augmentin tablet

INTERVENTIONS:
Drug: Augmentin tablet
  Other Names: Experimental: Augmentin; Augmentin 3 tablets (Amoxicilin:clavualanate=2:1) bid, for 14days

SUMMARY:
This study has an open-label, one-sequence, multiple drug administration design. The purpose of this study is as follows;

* To evaluate the change of liver function according to glutathione s-transferase (GST) genotype after the multiple administration of amoxicillin/clavulanate.
* To evaluate the intrinsic metabolite, human leukocyte antigen (HLA) genotype, and microRNA (miRNA) based on liver function change as the candidate biomarker for DILI.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with sufficient ability to understand the nature of the study and any hazards of participating in it. Provide written informed consent after being fully informed about the study procedures
2. Healthy male of female subjects aged 20 - 45 years
3. Subjects whose body mass index (BMI) in the range 18.5 kg/m2 (inclusive) - 27 kg/m2 (exclusive)

Exclusion Criteria:

1. Subject with clinically significant disease in liver, kidney, nerve system, respiratory system, endocrine system, blood, tumor, urinary system, cardiovascular system, mental disease or with medical history
2. Subject who has taken any prescribed drugs, herbal agents or crude drugs within 2 weeks before study drug administration
3. Subject who did blood donation during 1 months before the study or Blood donation during 2 months before the study
4. Subject with presence or history of severe adverse reaction to study drug
5. Subject who cannot prevent pregnancy during the study period.
6. Female subject who are pregnant.
7. Subject who drank over 21 units/week of alcohol or subjects who would not be able to stop drinking alcohol during the hospitalization
8. Subject who are Heavy smoker more than 10 cigarettes/day within 3 months prior to screening or subjects who would not be able to stop smoking during the hospitalization.
9. Subject judged not eligible for study participation by investigator.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Aspartate Aminotransferase (AST) | 22 days
Alanine Aminotransferase (ALT) | 22 days
Alkaline phosphatase (ALP) | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Jieon Lee, Seoul
  - Seoul National University Hospital, Seoul